CLINICAL TRIAL: NCT05413200
Title: Investigation of the Effect of Oral Isotretinoin on Clinical Severity, Skin Thickness, and Elasticity in Patients With Moderate to Severe Acne Vulgaris and Atrophic Acne Scar by Shear-Wave Elastography
Brief Title: Investigation of the Effect of Oral Isotretinoin on Skin Thickness and Elasticity in Patients With Atrophic Acne Scar
Status: Completed | Type: Observational
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Cemre Busra Turk, Principal Investigator, Istanbul Training and Research Hospital
Other Study IDs: 98
Record Dates: First submitted 2022-06-04; First posted 2022-06-09 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Acne Vulgaris; Isotretinoin; Atrophic Acne Scar
Keywords: acne vulgaris; oral isotretinoin theraphy; atrophic acne scars; Shear-Wave Elastography; skin elasticity
MeSH Terms: conditions — Acne Vulgaris | interventions — Isotretinoin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients diagnosed with moderate and severe AV accompanied by atrophic acne scars
  Interventions: Drug: Isotretinoin

INTERVENTIONS:
Drug: Isotretinoin — oral isotretinoin with a standard dose regime for 90 days

SUMMARY:
Acne scar is a common complication of acne vulgaris (AV). Early and effective treatment of AV has a crucial role in managing both acne and acne scarring. Oral isotretinoin (OI) is a widely preferred agent in treating moderate and severe AV worldwide. It has been shown that topical retinoids can also be effective in the treatment of atrophic acne scars. However, there is no study in the literature evaluating the effectiveness of OI protocol on atrophic scars with objective data. With the developing sonoelastography technology in recent years, a quantitative, objective, and reliable examination of the elasticity of the skin and subcutaneous tissue can be provided. In this study, for a detailed and objective evaluation of the effects of OI on atrophic acne scars, we investigate the AV severity, atrophic scar grade, scar size (SS), dermis and subcutaneous tissue thickness (STT), and changes in scar and subcutaneous tissue elastic modulus (EM) in moderate and severe AV patients with atrophic acne scars by clinical observation and SWE.

Materials and Methods: It was designed as a single-center, prospective and observational study. Ethics committee approval was obtained. Thirty patients who applied to the Istanbul Training and Research Hospital, Dermatology Department, between November 2021 and January 2022 diagnosed with moderate and severe AV accompanied by atrophic acne scars were included in the study. Demographic characteristics of the patients were recorded. We started the OI with a standard dose regime. On days 0 and 90 of treatment, each patient's AV and scar severity; were evaluated with the global acne grading system (GAGS) and the Goodman and Baron Qualitative Global Scar Rating System (GSRS). On the same days, the dermal thickness (DT), STT, SS, scar, and subcutaneous tissue EM on the right and left cheeks were measured by the same experienced radiologist with SWE. Appropriate statistical methods analyzed the results.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* Being under 65 years old
* Moderate to severe acne vulgaris with atrophic acne scars
* Absence of keloidal or hypertrophic scars
* Planning the use of oral isotretinoin in the treatment
* No additional disease
* Not smoking
* Consent to participate in the study and treatment

Exclusion Criteria:

* Using isotretinoin in the last 1 year
* Using topical or systemic medication in addition to oral isotretinoin for the treatment of acne vulgaris
* Having a keloidal or hypertrophic scar
* Being in pregnancy and lactation period
* To plan a pregnancy or are unable to adapt to contraception
* Known chronic diseases; skin cancer and other cancers, uncontrolled such as diabetes, hepatic failure/dysfunction, renal failure/dysfunction, neuromuscular diseases, autoimmune connective tissue diseases, hematological diseases, malabsorption diseases, inflammatory bowel diseases, pseudotumor cerebri, psychiatric diseases, and alcoholism.
* Severe hypercholesterolemia (>250 mg/dL), hypertriglyceridemia (> 500 mg/dL)
* Elevated liver function tests (ALT, AST, GGT, ALP) exceeding 3 times the upper limit
* Creatine kinase elevation exceeding 5 times the upper limit
* Using regular medication for another known disease
* To smoke
* A dermatological pathology other than facial acne vulgaris. (seborrheic dermatitis, rosacea, perioral dermatitis, herpes infection, impetigo, cutaneous lupus erythematosus, solar keratosis)
* Using Vitamin A
* Those who have or will receive a blood transfusion (during treatment or within 1 month after treatment)
* Hypersensitivity to the drug's preservatives
* Unrealistic expectations from treatment

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Thirty patients who applied to the Istanbul Training and Research Hospital, Dermatology Department, between November 2021 and January 2022 diagnosed with moderate and severe AV accompanied by atrophic acne scars were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-04-07 (Actual); Study Completion 2022-06-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline atrophic acne scar severity at 90 days | Day 0-90
  Change from baseline Goodman and Baron Qualitative Global Scar Rating System (first grade: grade 1, last grade: grade 4. Scar severity increases with increasing grade) at 90 days
Change from baseline skin thickness at 90 days | Day 0-90
  Change from baseline dermal and subcutaneous tissue thickness at 90 days
Change from baseline skin elasticity at 90 days | Day 0-90
  Change from baseline scar and subcutaneous tissue elasticity at 90 days

SECONDARY OUTCOMES:
Change from baseline acne vulgaris severity at 90 days | Day 0-90
  Change from baseline Global Acne Grading System (minimum score:0, maximum score: 44, severity increases with increasing score) at 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No